CLINICAL TRIAL: NCT04028856
Title: Cohort Study on Efficacy and Safety of Interferon Intermittent Treatment of Chronic Hepatitis B
Brief Title: Cohort Study of Efficacy and Safety of Interferon Intermittent Treatment of Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY019
Record Dates: First submitted 2019-07-20; First posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; interferon; intermittent; HBV; HBsAg; HBV DNA
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Interferons

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuous interferon treatment group: Patients with chronic hepatitis B treated with continuous interferon for 48 weeks
  Interventions: Drug: interferon
- Intermittent interferon treatment group: patients with chronic hepatitis B treated with intermittent interferon for 48 weeks, in which interferon therapy was intermittent for 3 months
  Interventions: Drug: interferon

INTERVENTIONS:
Drug: interferon — Chronic hepatitis B patients were treated with interferon for 48 weeks

SUMMARY:
This study was a retrospective clinical observational cohort study. All patients with chronic hepatitis B (CHB) whose HBsAg decreased by less than 10% were treated continuously with interferon in the Department of Hepatology, Beijing Ditan Hospital, Beijing Medical University, Beijing Capital University, 2008.10-2017.4. The total interferon treatment time of the enrolled subjects was 48 weeks. The subjects were randomly divided into the following two observation cohorts: 1) patients with chronic hepatitis B treated with continuous interferon for 48 weeks; 2) intermittent interferon For 48 weeks of treatment for patients with chronic hepatitis B, the interferon treatment interval was 3 months. HBV DNA content, HBsAg/anti-HBs, HBeAg/anti-HBe and biochemical markers, serum AFP and liver imaging (liver ultrasound) were collected before treatment (baseline) and during treatment. The primary outcome measure was the rate at which HBsAg disappeared at 48 weeks of treatment. The secondary evaluation index was the 48-week HBeAg seroconversion rate. To investigate the efficacy, influencing factors and safety of interferon intermittent treatment of chronic hepatitis B.

DETAILED DESCRIPTION:
This study was a retrospective clinical observational cohort study. All patients with chronic hepatitis B (CHB) whose HBsAg decreased by less than 10% were treated continuously with interferon in the Department of Hepatology, Beijing Ditan Hospital, Beijing Medical University, Beijing Capital University, 2008.10-2017.4. The total interferon treatment time of the enrolled subjects was 48 weeks. The subjects were randomly divided into the following two observation cohorts: 1) patients with chronic hepatitis B treated with continuous interferon for 48 weeks; 2) intermittent interferon For 48 weeks of treatment for patients with chronic hepatitis B, the interferon treatment interval was 3 months. HBV DNA content, HBsAg/anti-HBs, HBeAg/anti-HBe and biochemical markers, serum AFP and liver imaging (liver ultrasound) were collected before treatment (baseline) and during treatment. The primary outcome measure was the rate at which HBsAg disappeared at 48 weeks of treatment. The secondary evaluation index was the 48-week HBeAg seroconversion rate. To investigate the efficacy, influencing factors and safety of interferon intermittent treatment of chronic hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic hepatitis B meet the diagnostic criteria of China Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015)

Exclusion Criteria:

* coinfection with other viruses including HCV, HDV, and HIV;
* syphilis antibody positive;
* co-exist other liver diseases including alcoholic liver disease, metabolic liver disease, fatty liver, drug induce liver injury, and autoimmune liver disease;
* complication of cirrhosis or liver cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B (CHB) with a reduction in HBsAg of less than 10% were treated with interferon for 6 months. All patients with chronic hepatitis B were eligible for the diagnostic criteria of the Chinese Guidelines for the Prevention and Treatment of Chronic Hepatitis B (2015).
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of disappearance of HBsAg | after 48 weeks of treatment
  Rate of disappearance of HBsAg after 48 weeks of treatment

SECONDARY OUTCOMES:
HBeAg seroconversion rate | at the treatment of 48 weeks
  Treatment of 48 weeks HBeAg seroconversion rate

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Department of hepatology Division 2, Beijing Ditan Hospital, Capital Medical University
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li M, Xie S, Bi X, Sun F, Zeng Z, Deng W, Jiang T, Lin Y, Yang L, Lu Y, Zhang L, Yi W, Xie Y. An optimized mode of interferon intermittent therapy help improve HBsAg disappearance in chronic hepatitis B patients. Front Microbiol. 2022 Aug 30;13:960589. doi: 10.3389/fmicb.2022.960589. eCollection 2022. PMID 36110295